CLINICAL TRIAL: NCT04425512
Title: Delta Neutrophil Index and Neutrophil Lymphocyte Ratio in Differentiation of Thyroid Malignancy and Nodular Goiter
Brief Title: Delta Neutrophil Index and Neutrophil Lymphocyte Ratio in Thyroid Malignancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Mehmet Buğra Bozan, Professor, Assistant, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 355
Record Dates: First submitted 2020-04-23; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Thyroid Cancer; Thyroid Nodule; Thyroid Diseases; Delta Neutrophyl Index; Immature Granulocyte Count; Neutrophyl to Lymphocyte Ratio
Keywords: Delta neutrophyl index; Immature granulocyte count; Thyroid Cancer; Thyroid Nodule; Neutrophyl to lymphocyte ratio
MeSH Terms: conditions — Thyroid Neoplasms; Thyroid Nodule; Thyroid Diseases | interventions — Blood Cell Count

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Thyroid Malignancy (Active Comparator): Thyroidectomy
  Interventions: Diagnostic Test: Complete Blood Count
- Benign Thyroidal Goitor (Sham Comparator): Thyroidectomy
  Interventions: Diagnostic Test: Complete Blood Count
- Control Group (Other): Selective lichtenstein procedure for inguinal hernia
  Interventions: Diagnostic Test: Complete Blood Count

INTERVENTIONS:
Diagnostic Test: Complete Blood Count — Complete Blood Count samples
  Other Names: Thyroidectomy

SUMMARY:
Thyroid surgery is the most common surgical procedure among endocrine surgeries. It is performed in patients with suspected malignancy, patients diagnosed with malignancy, and for toxic nodular goiter [1]. Fine-needle aspiration biopsy (FNAB) is used as a daily technique in preoperative evaluation to differentiate malignant and benign nodules. However, complications including hematoma formation, tumor transplantation along the needle trace, thyroid nodule infarction and vascular proliferation can be seen even in this minimally invasive procedure [2]. Therefore, the differentiation of benign and malignant groups using non-interventional methods before surgery has become important.

Cancer-related inflammation, including papillary thyroid carcinoma, is involved in carcinogenesis and progression of neoplastic disease [3,4]. Neutrophils induced by the tumor can accelerate tumor metastasis [3,5]. Lymphocytes, as the cornerstone of the adaptive immune system, inhibit tumor cell proliferation and migration as well as destroying metastases [3,6]. Previous studies have shown that increased lymphocyte count has a positive effect on better survival in patients with advanced cancer [7]. Furthermore, Kupffer cells, also known as liver macrophages, destroy circulating cancer cells and help the distribution of tumor cells via circulation. Therefore, routine blood tests have been investigated as a predictive or prognostic factor for carcinomas since blood parameters in these tests show whether there is inflammation. Neutrophil count, lymphocyte count, neutrophil-lymphocyte ratio (NLR), lymphocyte-monocyte ratio (LMR), mean platelet volume (MPV), and platelet distribution width (PDW) have been studied in terms of numerous malignancies [3].

Tumor-related inflammation is activated the bone marrow and inflammation induced by malignancies. Inflammatory activity that is poorly controlled or uncontrollable may be responsible for malignant transformation [8]. At this point, NLR has previously been shown to be useful in the differentiation of thyroid malignancies and benign thyroid diseases [9]. Delta neutrophil index (DNI) / increased number of immature granulocytes (IG) represents active bone marrow. Delta neutrophil index, which is manifested by IG formation in inflammatory and infectious events, shows changes in the white blood cell count [10].

This study aimed to evaluate the relation between the automatically calculated DNI/IG count and manually calculated NLR from the preoperative complete blood count (CB) parameters, and thyroid malignancies with a cost-effective non-invasive method before surgery or biopsy as the indicator of the malignant inflammatory response in the differentiation of nodular goiter and thyroid malignancy.

DETAILED DESCRIPTION:
Material-Methods Patients over the age of 18 who underwent thyroid surgery and who were operated on non-malignant benign causes (inguinal hernia) under selective conditions without any thyroid disease between November 2014 and November 2019 in Kahramanmaraş Sütçü İmam University Department of General Surgery were evaluated in this retrospective case-control cohort study. Patients in the thyroid pathology group (Group T) were divided into two subgroups according to their pathologic results: malignant (Group M) and benign thyroid disorders (Group B). Patients operated for inguinal hernia, were selected as control group (Group C).

All procedures performed in studies involving human participants were in accordance with the ethical standards of the institutional and/or national research committee and with the 1964 Helsinki declaration and its later amendments or comparable ethical standards.

Preoperative biopsy results of patients undergoing FNAB in the preoperative period were investigated according to the Bethesda Classification System [11]. Neutrophil - lymphocyte count in the routine complete blood count (CBC) values, which were measured in the preoperative period and the postoperative sixth-month follow-ups, were recorded retrospectively and calculated manually. DNI (IG percentage) and IG counts were recorded from the values measured automatically in the CBC performed in the preoperative period and the postoperative sixth-month. Patient data were obtained from patient epicrisis forms and preoperative laboratory and postoperative pathology results recorded in the computer system.

Statistical Analysis The power analysis of the study was conducted with G-Power 3.0.10 programming system. Estimated power analysis and the sample size with an 0.8 power and effect size 0.1 according to three groups evaluation for 2 repeated measures in need of total 246 samples.

Statistical analysis was performed using IBM Social Package for the Social Sciences (SPSS) version 20 software. In the evaluation of independent groups, Kolmogorov-Smirnov and Shapiro-Wilk tests were used to determine if the distrubiton of variables were normal or not. Student t-test or Mann-Whitney U test was used to evaluate the numerical data between Group C and Group T. ANOVA or Kruskal Wallis test was used to evaluate numerical data for subgroup relations with Group C. Chi-square test or Fischer's exact test was used to evaluate categorical data. The repeated-measures ANOVA was used to evaluate the differences between the preoperative and postoperative periods. The data were evaluated using Posthoc Tukey's B test following the variance analysis. Sensitivity and specificity values and cut-off values were obtained via the receiver operating characteristic (ROC) analysis to evaluate the effectiveness of NLR, IG count, and DNI.

Numerical data were expressed as mean ± standard deviation (minimum-maximum values) or median (minimum-maximum values) according to the normal distribution. Categorical values were expressed as percentages (%).

ELIGIBILITY:
Inclusion Criterias:

* Operated thyroid malignancy patients (Total thyrodectomy, complementary thyroidectomy)
* Operated benign thyoridal goitor patients
* Selectively operated inguinal hernia patients without any concomitant malignancy
* Selectively operated inguinal hernia patients without any thyroid disorder

Exclusion Criterias:

* Patients undergoing emergent surgery
* Patients with concomitant rheumatologic disease undergoing thyroid surgery in selective conditions
* Patients with concomitant rheumatologic disease undergoing inguinal hernia operation in selective conditions
* Patients with concomitant thyroid disease undergoing inguinal hernia operation in selective conditions
* Patients with concomitant any malignancy undergoing inguinal hernia operation in selective conditions
* Patients whose data were not available or were missing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 333 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Delta neutrophyl index for thyroid malignancies | retrospective 5 year
  The correlation between DNI and thyroid cancer
Immature granulocyte count for thyroid malignancies | retrospective 5 year
  The correlation between DNI and thyroid cancer
Neutrophyl to lymphocyte ratio for thyroid malignancies | retrospective 5 year
  The correlation between DNI and thyroid cancer

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith PW, Hanks LR, Salomonev LJ, Hanks JB. Sabiston's Text Book of Surgery 20th Edition, The Biological Basis of Modern Surgical Practice. 20th edition, Philedelphia/USA: Elsevier; 2017. Chapter 36 Thyroid. Pp: 881-922
- [Background] Madden LL, Nagatsuka M, Vasi AZ, Madrecha J, Smith LJ. Nerve Injury During Ultrasound-Guided Thyroid Biopsy-A First Reported Complication of Permanent Vocal Fold Paralysis. Ear Nose Throat J. 2021 Sep;100(5_suppl):663S-666S. doi: 10.1177/0145561320902855. Epub 2020 Feb 10. PMID 32041420
- [Background] Wen W, Wu P, Li J, Wang H, Sun J, Chen H. Predictive values of the selected inflammatory index in elderly patients with papillary thyroid cancer. J Transl Med. 2018 Sep 21;16(1):261. doi: 10.1186/s12967-018-1636-y. PMID 30241494
- [Background] Balkwill F, Mantovani A. Inflammation and cancer: back to Virchow? Lancet. 2001 Feb 17;357(9255):539-45. doi: 10.1016/S0140-6736(00)04046-0. PMID 11229684
- [Background] Coffelt SB, Wellenstein MD, de Visser KE. Neutrophils in cancer: neutral no more. Nat Rev Cancer. 2016 Jul;16(7):431-46. doi: 10.1038/nrc.2016.52. Epub 2016 Jun 10. PMID 27282249
- [Background] Bastid J, Bonnefoy N, Eliaou JF, Bensussan A. Lymphocyte-derived interleukin-17A adds another brick in the wall of inflammation-induced breast carcinogenesis. Oncoimmunology. 2014 Mar 27;3:e28273. doi: 10.4161/onci.28273. eCollection 2014. PMID 25050201
- [Background] He JR, Shen GP, Ren ZF, Qin H, Cui C, Zhang Y, Zeng YX, Jia WH. Pretreatment levels of peripheral neutrophils and lymphocytes as independent prognostic factors in patients with nasopharyngeal carcinoma. Head Neck. 2012 Dec;34(12):1769-76. doi: 10.1002/hed.22008. Epub 2012 Feb 9. PMID 22318781
- [Background] Lee F, Yang PS, Chien MN, Lee JJ, Leung CH, Cheng SP. An Increased Neutrophil-to-Lymphocyte Ratio Predicts Incomplete Response to Therapy in Differentiated Thyroid Cancer. Int J Med Sci. 2018 Nov 23;15(14):1757-1763. doi: 10.7150/ijms.28498. eCollection 2018. PMID 30588200
- [Background] Kocer D, Karakukcu C, Karaman H, Gokay F, Bayram F. May the neutrophil/lymphocyte ratio be a predictor in the differentiation of different thyroid disorders? Asian Pac J Cancer Prev. 2015;16(9):3875-9. doi: 10.7314/apjcp.2015.16.9.3875. PMID 25987053
- [Background] Kim TY, Kim SJ, Kim YS, Lee JW, Park EJ, Lee SJ, Lee KJ, Cha YS. Delta neutrophil index as an early predictive marker of severe acute pancreatitis in the emergency department. United European Gastroenterol J. 2019 May;7(4):488-495. doi: 10.1177/2050640619838359. Epub 2019 Mar 14. PMID 31065366
- [Background] Cibas ES, Ali SZ. The 2017 Bethesda System for Reporting Thyroid Cytopathology. Thyroid. 2017 Nov;27(11):1341-1346. doi: 10.1089/thy.2017.0500. PMID 29091573